CLINICAL TRIAL: NCT04975087
Title: Reliability, Validity, and Cross-cultural Adaptation of the Turkish Version of the Profile of Fatigue and Discomfort - Sicca Symptoms Inventory in Sjogren Patients
Brief Title: The Profile of Fatigue and Discomfort - Sicca Symptoms Inventory
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fulden Sarı, research assistant, Gazi University
Other Study IDs: 206
Record Dates: First submitted 2021-07-15; First posted 2021-07-23 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Primary Sjögren's Syndrome
Keywords: sjogren; validity; reliability; fatigue; sicca symptoms
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients group: Individuals with primary Sjögren's syndrome
  Interventions: Other: Patients group

INTERVENTIONS:
Other: Patients group — Patients will complete the mentioned questionnaires.

SUMMARY:
Primary Sjögren's syndrome (pSS) is a chronic, systemic autoimmune disease characterized by disorders of the lacrimal and salivary glands. The disease can be seen in systemic involvement by affecting any organ. It may result in skin, lung and kidney involvement as well as symptoms such as vasculitis and neuropathy. Patients with PSS often report fatigue as an important symptom to manage. Fatigue, defined as an overwhelming feeling of fatigue, lack of energy, and exhaustion, is associated with poor health and functional impairment.

Fatigue is a common symptom of pSS. This symptom is the most important cause of loss of function in patients. It is thought that as a result of fatigue in pSS, decrease in mental health related to physical activity level and quality of life in patients, sleep problems, depression and loss of ability to work. Several mechanisms have been proposed to explain the occurrence of fatigue among sjogren patients, but its underlying physiological basis has not been adequately defined. Therefore, it is a complex, multifaceted and poorly understood symptom.

In population-based studies, approximately 20% of healthy adults report experiencing fatigue, and this rate rises to 60%-70% among patients with autoimmune disorders. Fatigue is the most common non-exocrine symptom in pSS, and the prevalence of fatigue disability among patients with pSS has been reported to be approximately 70%.

DETAILED DESCRIPTION:
In order to evaluate fatigue in primary Sjögren's syndrome patients, questionnaires such as FACIT Fatigue Scale, Sjögren's Syndrome EULAR Patient Reporting Index, Fatigue Severity Scale, Fatigue Multidimensional Assessment Scale and Short Form-36, which are also used in many disease groups, are used. Although the importance of the effect of fatigue on pSS patients has been demonstrated in studies, most of the fatigue assessment questionnaires used are not pSS specific. For this reason, Bowman et al. They developed the Fatigue and Discomfort Profile - Sikka Symptoms Scale (PROFAD-SSI) to assess multidimensional fatigue in patients with pSS, considering disease symptoms. PROFAD-SSI is scored from 0 to 7 on an 8-point Likert scale. The 19-item scale evaluates patients in 8 different dimensions: somatic fatigue, mental fatigue, arthralgia, vascular dysfunction, oral dryness, ocular dryness, cutaneous and vaginal dryness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary Sjögren's syndrome
* Patients between the ages of 18-65
* Being literate

Exclusion Criteria:

* Having cognitive disorders
* Having another rheumatological diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary Sjögren's syndrome between the ages of 18-85
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
the Profile of Fatigue and Discomfort - Sicca Symptoms Inventory | 10 minutes
  It is scored between 0-7 on an 8-point Likert scale. The 19-item scale evaluates patients in 8 different dimensions: somatic fatigue, mental fatigue, arthralgia, vascular dysfunction, oral dryness, ocular dryness, cutaneous and vaginal dryness.

CONTACTS AND LOCATIONS:
Overall Officials: Deran OSKAY, Prof, Study Director — Gazi University
Locations (1):
- Gazi University, Çankaya, Ankara, Turkey (Türkiye)